CLINICAL TRIAL: NCT04911283
Title: Mehmet Akif İnan Education and Research Hospital
Brief Title: Brucella Serology and History of Brucellosis in Patients With Modic Changes Type 1
Status: Completed | Type: Observational
Sponsor: Veysel Delen (Other)
Responsible Party: Sponsor-Investigator, Veysel Delen, Department of Physical Medicine and Rehabilitation, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Organization: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Other Study IDs: SUEADH
Record Dates: First submitted 2021-05-25; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Brucellosis; Spinal Degeneration
MeSH Terms: conditions — Brucellosis | interventions — Health Records, Personal; Pyrin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MCs type 1 patients (study group; n=37)
  Interventions: Other: Brucella serology test; Other: Medical history for brucellosis
- MCs type 2 patients (comparator group; n=44)
  Interventions: Other: Brucella serology test; Other: Medical history for brucellosis
- healthy controls (n=37)
  Interventions: Other: Medical history for brucellosis

INTERVENTIONS:
Other: Brucella serology test — MCs type 1 and type 2 patients were examined in terms of Brucella serology by using agglutination with Coombs test.
  Groups: MCs type 1 patients (study group; n=37); MCs type 2 patients (comparator group; n=44)
Other: Medical history for brucellosis — Both of the MCs groups and healthy controls were investigated for their medical history regarding brucellosis.

SUMMARY:
Objective: This study aims to examine Brucella serology and history of brucellosis in patients with lumbar Modic changes (MCs) type 1, considering results from cross-sectional and case-control comparisons.

Design: In comparative cross-sectional design, MCs type 1 patients (study group) and MCs type 2 patients (comparator group) were examined in terms of Brucella serology by using agglutination with Coombs test. In addition, in comparative case-control design, both of the MCs groups and age/sex-matched healthy controls were investigated for their medical history regarding brucellosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar Modic changes type 1
* Patients with lumbar Modic changes type 2
* Participant who given informed consent for the study

Exclusion Criteria:

* Patients aged<18 years
* History of serious lumbar trauma
* Lumbar spinal surgery
* Scoliosis
* Cooperation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with MCs and age/sex-matched healthy controls
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Serology for brucellosis | 30 minutes
History of brucellosis | 7 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Veysel Delen, Principal Investigator — Mehmet Akif İnan Hospital
Locations (1):
- Mehmet Akif İnan Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No